CLINICAL TRIAL: NCT06843551
Title: A Phase 2 Single Arm Trial of Stereotactic Body Radiation Therapy Followed by Dual Immune Checkpoint Inhibition for Patients With Metastatic Pancreatic Ductal Adenocarcinoma - The Miami "EMPIRE" Trial - Eradication of Metastatic Pancreatic Cancer With Immuno-Radiation
Brief Title: The Miami "EMPIRE" Trial - Eradication of Metastatic Pancreatic Cancer With Immuno-Radiation
Acronym: EMPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Benjamin Spieler (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor-Investigator, Benjamin Spieler, Assistant Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240455
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation, Botensilimab Combined with Balstilimab Treatment Group (Experimental): Participants in this group will receive Stereotactic Body Radiation Therapy (SBRT), followed by Botensilimab immunotherapy (ImT) for up to 24 weeks, in combination with Balstilimab ImT for up to one year.
  Total participation duration is up to five years.
  Interventions: Radiation: Stereotactic Body Radiation Therapy; Drug: Botensilimab; Drug: Balstilimab

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — The radiation therapy (RT) prescription biologically effective dose (BED10) goal for tumor (α/β=10) aims to achieve at least BED10= 60 Gy for a single fraction plan and at least BED10=100 Gy for a multi-fraction plan. This equates to a prescription dose of at least 20 Gy in a single fraction, 42 Gy over 3 fractions, 50 Gy over 5 fractions, and 62 Gy over 10 fractions.
  Radiation therapy must be completed for up to 10 daily treatments within a 15-day course.
Drug: Botensilimab — Participants will be receive 75mg of Botensilimab immunotherapy administered via intravenous infusion, every six weeks for up to 4 doses, about 24 weeks. Botensilimab therapy will begin no later than seven (7) days after completion of radiation therapy.
Drug: Balstilimab — Participants will receive 240mg of Balstilimab immunotherapy, administered via intravenous infusion, every 2 weeks for up to one (1) year. Balstilimab therapy will begin no later than seven (7) days after completion of radiation therapy.

SUMMARY:
The purpose of this study is to assess if radiation therapy (which uses high-energy radiation to damage or destroy cancer cells) combined with immune checkpoint inhibitors (medications that helps the body recognize and attack cancer cells) will be beneficial for patients with metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Histologically or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma.
3. Microsatellite stable (MSS) disease by pathologic assessment.
4. Patients must have measurable disease as defined by RECIST 1.1.
5. Progression on ≥1 line of systemic therapy.
6. No concomitant therapy with any of the following: interleukin (IL)-2, interferon, non study immunotherapy regimens, cytotoxic chemotherapy, immunosuppressive agents, other investigational therapies, and/or chronic use of systemic corticosteroids.
7. No known infection with human immunodeficiency virus (HIV) or active infection with Hepatitis B.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
9. Life expectancy ≥3 months.
10. Patients must have the following lab values obtained <4 weeks prior to starting protocol treatment:

    1. absolute neutrophil count (ANC) ≥1,000 cells/μL
    2. white blood count (WBC) ≥2,000 cells/μL
    3. platelets ≥75,000 per μL
    4. hemoglobin ≥8.0 g/dL
    5. creatinine clearance ≥40 mL/min)
    6. serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
    7. aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤3 × ULN (or ≤5 × ULN in patients with liver metastases)
    8. international normalized ratio or prothrombin time ≤1.5 × ULN
    9. activated partial thromboplastin time ≤2.5 × ULN
    10. absolute lymphocyte count (ALC) ≥1000 cells/μL at baseline
11. At least 1 previously unirradiated lesion amenable to pre-treatment biopsy.
12. No limit on overall numbers of lesions, but liver tumor burden ≤25% of total liver volume.
13. Women of childbearing potential (WOCBP): negative serum pregnancy test (within 7 days prior to Day 1 of protocol therapy)

    a. Females of non-childbearing potential are defined as: i. ≥ 50 years of age and has not had menses for greater than 1 year ii. Amenorrheic for ≥ 2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation iii. Status is post-hysterectomy, bilateral oophorectomy, or tubal ligation.
14. Male and female patients of reproductive potential must use effective methods of contraception or abstain from sexual activity for the course of the study through at least 6 months after the last dose of balstilimab and/or botensilimab. See Section 4.11, Contraception.

Exclusion Criteria:

1. Liver tumor burden exceeding 25% of total liver volume.
2. Active, untreated central nervous system (CNS) metastases.
3. Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years of the start of study treatment (i.e., with use of disease-modifying agents or immunosuppressive drugs).
4. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses (≤ 10 mg daily prednisone equivalent) are permitted in the absence of active autoimmune disease.
5. Previous external beam radiation therapy to the liver or radioisotope therapy directed to the liver or any liver embolization.
6. Clinically significant ascites requiring a paracentesis in the last 4 weeks, or clinically significant history of liver failure defined as any prior episode of hepatic encephalopathy and/or any prior history of an elevated serum ammonia level.
7. Partial or complete bowel obstruction within the last 3 months prior to study enrollment, signs/symptoms of bowel obstruction, or known radiologic evidence of impending obstruction.
8. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of study enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication.

   a. QT interval corrected using Fridericia's formula (QTcF) of > 480 ms.
9. Prior allogeneic organ transplantation.
10. Treatment with chemotherapy or targeted therapy within 2 weeks prior to initiating EMPIRE treatment.
11. Persistent grade ≥2 adverse events (aEs) from prior therapy (except neuropathy).
12. Known additional malignancy requiring active treatment.
13. History of non-infectious pneumonitis.
14. Active infection requiring antibiotic.
15. Live vaccine within 30 days of protocol treatment.
16. Severe acute respiratory syndrome (SARS) coronavirus 2 (CoV 2) (SARS-CoV-2) vaccine or booster < 7 days before Cycle 1 Day 1 (C1D1). For vaccines requiring more than 1 dose, the full series should be completed prior to C1D1, when feasible. Booster shot not required but also must be administered > 7 days from C1D1 or > 7 days from future cycle on study.
17. History of severe hypersensitivity reaction to monoclonal antibody.
18. Participants with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | Up to 15 months
  The Clinical Benefit Rate (CBR) among participants will be reported. CBR is the number of participants achieving complete response (CR), partial response (PR) or stable disease after start of study therapy. Response will be assessed using Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) 1.1 criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 15 months
  Objective response rate will be reported, based on best response according to Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) 1.1 criteria. Objective response (OR) is defined as the number of participants with confirmed complete response (CR) or confirmed partial response (PR) to study therapy.
Progression-Free Survival (PFS) | Up to 5 years
  Progression-free survival (PFS) among participants will be reported. PFS is defined as the elapsed time in months since the start of radiation therapy until the first documentation of disease progression or death.
Overall Survival (OS) | Up to 5 years
  Overall survival (OS) among participants will be reported. OS is defined as the elapsed time in months from the start of radiation therapy until death by any cause.
Number of Participants Experiencing Grade 3 or Higher Toxicities | Up to 15 months
  The number of participants experiencing Grade 3 or higher toxicities will be reported using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Spieler, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No